CLINICAL TRIAL: NCT04625881
Title: Effects of an Apple Derived Fibre Supplement on Digestive Symptoms and Evacuation Frequency in People With Constipation
Brief Title: Effects of an Apple Derived Fibre Supplement on Constipation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Collaborators: Gladys Barrera Acevedo (Unknown)
Responsible Party: Principal Investigator, Daniel Bunout, Full professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Manzana
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Constipation; Functional Gastrointestinal Disorders
Keywords: constipation; dyspepsia
MeSH Terms: conditions — Constipation; Gastrointestinal Diseases; Dyspepsia

STUDY DESIGN:
Intervention Model Description: Double blind parallel study comparing a fiber supplement with a fiberless placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active product and placebo will have the same appearance. All vials will have an unique numerical code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active product (Active Comparator): A powder containing 20 g of apple derived fiber will be consumed daily
  Interventions: Dietary Supplement: Apple derived fiber
- Placebo (Placebo Comparator): A rice derived placebo devoid of fiber and aromatized with apple fragancy will be provided
  Interventions: Dietary Supplement: Apple derived fiber

INTERVENTIONS:
Dietary Supplement: Apple derived fiber — This is a combination of soluble and insoluble fiber

SUMMARY:
We will conduct a 2 months clinical intervention in which a 20 g appled derived fibre supplement will be compared with a placebo without fibre. The main outcome will be the reduction in the Gastrointestinal System Rating Scale

DETAILED DESCRIPTION:
Participants with constipation and mild gastrointestinal symptoms will be invited to participate. Those with alarming symptoms such as gastrointestinal bleeding or weight loss, those using laxatives or medications with anticholinergic actions will be excluded from the study At baseline, participants will be weighed and interrogated about Their gastrointestinal symptoms using the "Gastrointestinal symptom rating scale" Their type of stools using the Bristol visual stool scale The number of complete spontaneous bowel movements per week Afterwards, they will be randomized, balancing by age, gender and body mass index to receive in a doubly blind fashion A 20 g/day powder with apple derived fiber A similarly looking placebo powder The intervention will last 8 weeks. Every two weeks, participants will be cited to provide a new supply of the product, retrieve the used vials and be interrogated using the same tools as baseline. At the end of the intervention, participants will be weighed again

ELIGIBILITY:
Inclusion Criteria:

* presence of constipation or functional gastrointestinal symptoms

Exclusion Criteria:

having serious cardiovascular, kidney or hepatic diseases

* gastrointestinal bleeding weight loss use of laxatives use of medications with anticholinergic actions

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal symptom rating scale | every 2 weeks during 8 weeks
  This scale assesses abdominal pain, bloating and type of stools

SECONDARY OUTCOMES:
Number of complete spontaneous bowel movements per week | every 2 weeks during 8 weeks
  the title is auto-explicative

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Nutrition and Food Technology University of Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided
All information will be in databases without any identification information of participants

REFERENCES:
- [Result] Wiklund IK, Fullerton S, Hawkey CJ, Jones RH, Longstreth GF, Mayer EA, Peacock RA, Wilson IK, Naesdal J. An irritable bowel syndrome-specific symptom questionnaire: development and validation. Scand J Gastroenterol. 2003 Sep;38(9):947-54. doi: 10.1080/00365520310004209. PMID 14531531
- [Result] Liu Z, Yan S, Wu J, He L, Li N, Dong G, Fang J, Fu W, Fu L, Sun J, Wang L, Wang S, Yang J, Zhang H, Zhang J, Zhao J, Zhou W, Zhou Z, Ai Y, Zhou K, Liu J, Xu H, Cai Y, Liu B. Acupuncture for Chronic Severe Functional Constipation: A Randomized Trial. Ann Intern Med. 2016 Dec 6;165(11):761-769. doi: 10.7326/M15-3118. Epub 2016 Sep 13. PMID 27618593